CLINICAL TRIAL: NCT06223191
Title: Comparing Brief Negotiated Interview, Narrative Interview, and Standard Care to Reduce Readmission: A 2024 Clinical Trial in Substance Use Disorder Patients at Santa Rosita Psychiatric Specialties Hospital
Brief Title: Reducing Readmissions: BNI Trial in Substance Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Principal Investigator, Carlos Manuel Rosales Gomez, Principal Investigator, Universidad Nacional Autonoma de Honduras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BNIReadmissions
Record Dates: First submitted 2023-12-21; First posted 2024-01-25 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Substance Use Disorders; Substance Withdrawal
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief Negotiated Interview (Experimental): The BNI helps health care providers explore health behavior change with patients in a respectful, non-judgmental way within a finite time period. Instead of telling the patient what changes he/she should make, the BNI is intentionally designed to elicit reasons for change and action steps from the patient. It gives the patient voice and choice, making any potential behavior changes all the more empowering to the patient.
  Interventions: Other: Brief Negotiated Interview
- Narrative Interview (Placebo Comparator): The Narrative Interview is a therapeutic approach that aims to motivate the individual's conscious and transformative knowledge, skills, and capabilities. This interview is based on the technical components of narrative therapy, where the patient narrates their story, using externalizing language and considering social and political aspects related to the issue. It will focus on exploring past and present feelings, thoughts, and actions.
  Interventions: Other: Narrative Interview
- Standards of Care (No Intervention): This arm includes the use of benzodiazepines (Diazepam or Lorazepam) when CIWA-Ar scale is ≥9. Other medications may include Thiamine, Potassium Chloride, oral rehydration salts, parenteral fluids, antiemetics, and gastric protectants if medically necessary. Patients undergo a psychological evaluation on the third day of admission. All patients receive at least one psychoeducational session on alcohol and substance use during their hospitalization. Psychiatric evaluation is available for those with dual diagnoses such as mood disorders, anxiety disorders, psychotic disorders, or multiple substance use. The total hospitalization time in the ward is 8 days.

INTERVENTIONS:
Other: Brief Negotiated Interview — The BNI is a specialized "brief intervention" for the medical setting, has foundations in motivational interviewing techniques. The BNI helps health care providers explore health behavior change with patients in a respectful, non-judgmental way within a finite time period. The BNI is in the form of an algorithm, or "script", that guides providers through the health intervention with carefully phrased key questions and responses, all at the providers' fingertips
  Arms: Brief Negotiated Interview
Other: Narrative Interview — The Narrative Interview is a therapeutic approach that aims to motivate the individual's conscious and transformative knowledge, skills, and capabilities. This interview is based on the technical components of narrative therapy, where the patient narrates their story, using externalizing language and considering social and political aspects related to the issue. It will focus on exploring past and present feelings, thoughts, and actions.
  Arms: Narrative Interview

SUMMARY:
The aim of this clinical trial is to assess the effectiveness of Brief Negotiated Interview (BNI) in comparison to Narrative Therapy and Standard Care in reducing readmissions among male patients aged 18 and above with a history of substance use disorder The main questions it aims to answer is: Does the Brief Negotiated Interview reduces rehospitalization rates at least to 50%? Participants will be submitted to a Structured interview with motivational interviewing techniques. Researchers will compare 2 control groups one with standards of care and the other one with a narrative interview to see if they reduce readmission.

DETAILED DESCRIPTION:
The research investigates the effectiveness of the Brief Negotiated Interview (BNI) compared to Narrative Interview and Standards of Care in reducing readmissions among patients with Substance Use Disorder (SUD) in the Alcoholic Detoxification Unit of Santa Rosita Psychiatric Specialties Hospital in 2024. Employing a randomized clinical trial design, the study aims to address a critical gap in understanding the optimal intervention for this vulnerable population.

Study Design: This trial adopts a prospective, randomized, three-arm design, with participants randomly assigned to one of three groups: BNI, Narrative Interview, or Standard Care. The randomization process utilizes a computer-generated list, ensuring an allocation ratio of 1:1:1. The trial encompasses a recruitment period of three months, followed by a three-month follow-up period.

Participants: The target population comprises 150 male patients aged 18 or older admitted to the Alcoholic Detoxification Unit during January 2024.

Interventions:

Brief Negotiated Interview (BNI): Modeled after motivational interviewing techniques, BNI aims to empower patients to explore reasons for change. Administered as a single 30-minute session, BNI encourages patient autonomy in decision-making regarding behavioral changes related to substance use.

Narrative Interview: A 20-minute session applying narrative therapy techniques, encouraging patients to explore and reframe their stories concerning substance use. The session emphasizes externalizing issues and examining social and political factors contributing to the problem.

Standard Care: Following the Alcohol Detoxification Management Protocol, standard care includes pharmacological interventions (benzodiazepines, thiamine, etc.), psychological evaluation on the third day, psychoeducational sessions, and psychiatric assessment for dual diagnoses.

Outcomes: Primary outcomes involve measuring rehospitalization rates at three months, time to relapse, reduction in substance consumption, and changes in depressive and anxious symptoms.

Statistical Analysis:Descriptive statistics will characterize nominal and categorical variables. For continuous variables, means and standard deviations will be calculated. Chi-square tests will assess the relationship between rehospitalization and intervention groups. Risk ratios and incidence rates will be computed to determine the relative risk of readmission.

Ethical Considerations: The study adheres to CONSORT guidelines, receiving approval from the Institutional Review Board. Informed consent is obtained from all participants, ensuring comprehension of the study's purpose, risks, and benefits. Confidentiality is maintained, and participants are informed of their right to withdraw without interference in their clinical care.

Conclusion: This comprehensive research design integrates rigorous methodology, ethical considerations, and a tailored intervention approach to address the multifaceted challenges faced by patients with SUD. The outcomes are expected to contribute valuable insights to the field, guiding evidence-based practices for enhanced patient outcomes and reduced readmission rates

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 or older who are hospitalized in the Alcohol Detoxification Unit during the period of January to March of 2024
* Patients with a score on the AUDIT scale greater than 15.
* Patients with a score equal to or greater than 4 for any substance on the World Health Organization-ASSIST.
* Patients from the Alcohol Detoxification Unit who provide their consent to participate in the study.

Exclusion Criteria:

* Patients with a score on the AUDIT scale less than 15.
* Patients with a score on the WHO-ASSIST scale for substances less than 4.
* Patients from the Alcohol Detoxification Unit who do not provide their consent to participate in the study.
* Patients from the Alcohol Detoxification Unit diagnosed with Delirium Tremens, Acute Intoxication of any substance, or conditions that alter consciousness.
* Patients from the Alcohol Detoxification Unit diagnosed with intellectual disability documented in the medical records.
* Female patients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Hospital Readmission Rate | 3 months
  Measurement of the readmissions rate at 3 months from the study's initiation. This could be a key indicator to assess the impact of interventions on relapse prevention.
Risk Rate of Readmission | 3 months
  Measurement of the risk rate through the ratio of the readmission rate treatment group and the control group rate

SECONDARY OUTCOMES:
HADS Score | 3 months
  Assessment of the presence of depressive and anxious symptoms in patients with substance use. Through HADS ScaleThis primary outcome would directly address the participants' mental health as a result of the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M. Rosales, MD, Principal Investigator — Universidad Nacional Autonoma de Honduras
Locations (1):
- Facultad de Ciencias Medicas, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No